CLINICAL TRIAL: NCT00723814
Title: Blood Pressure Monitor Clinical Test
Status: Completed | Type: Observational
Sponsor: Andon Health Co., Ltd (Industry)
Other Study IDs: andonhealth
Record Dates: First submitted 2008-07-27; First posted 2008-07-29 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Blood Pressure
Keywords: normal

SUMMARY:
To monitor the blood pressure level of the patient

ELIGIBILITY:
Inclusion Criteria:

- IEC 60601-1-2

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult

PRIMARY OUTCOMES:
monitor the diastolic and systolic | 1 month